CLINICAL TRIAL: NCT00348049
Title: A Prospective, Randomized Trial Evaluating the Operational Efficacy of LASIK vs. PRK for the Correction of Low and Moderate Myopia in the Singapore Armed Forces
Brief Title: Efficacy of LASIK Versus PRK in Asians With Mild and Moderate Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Armed Forces (Unknown); Defence Medical Environmental Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R277/21/2002
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2002-10

CONDITIONS: Myopia
Keywords: LASIK; PRK; Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ; Photorefractive Keratectomy

INTERVENTIONS:
Procedure: Laser in Situ Keratomileusis (LASIK)
Procedure: Photorefractive Keratectomy (PRK)

SUMMARY:
Laser in situ keratomileusis (LASIK) and photorefractive keratectomy (PRK) are currently the 2 main refractive surgeries to correct myopia which are being performed worldwide, with more patients preferring LASIK to PRK because of better comfort and faster rehabilitation. However, in post-LASIK patients, there is a low risk of flap dislodgement. This risk increases with certain occupations which have a higher risk of trauma. Hence, there may be a role for PRK for people which such occupations, e.g. soldiers, parachutists, sportsman.

There are several non-randomised studies which show that PRK is as efficacious, predictable and safe as LASIK for low to moderate myopes. But there have been only a few randomized controlled studies to compare the efficacy and safety of the 2 treatment modalities and all studies comparing LASIK and PRK suffer from a high dropout rate during the follow-up period. We compared the efficacy, predictability, stability and safety of LASIK versus PRK over a one year duration with almost 100% attendance during all follow-up visits.

DETAILED DESCRIPTION:
This study is a prospective, randomized, clinical trial comparing the efficacy, predictability, stability and safety of LASIK versus PRK in a volunteer group of myopic military servicemen recruited from the Singapore Armed Forces. 132 subjects who were eligible for the study were randomized to undergo either LASIK or PRK in both eyes in a 2:1 ratio. 45 subjects (90 eyes) underwent PRK and 87 subjects (174 eyes) underwent LASIK.

An additional 59 subject underwent a non-randomised arm of the study and underwent PRK.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects were eligible for the study if they were 18 years old or older and had given informed consent; had stable myopia ranging from -2.00 to -5.00D of spherical equivalent myopia, but less than 2.00D of refractive astigmatism as determined by manifest refraction for at least 6 months; a best corrected visual acuity of at least 20/20 and a stable keratometry after not wearing soft contact lenses for at least 2 weeks and hard lenses for at least 3 weeks. Study subjects were required to have a minimum cornea thickness of at least 460um as measured by Orbscan pachymetry.

Exclusion Criteria:

* Subjects were excluded if they had corneal or anterior segment pathology, or myopic peripheral retinal degeneration or myopic macular degeneration; clinical signs of progressive or unstable myopia or keratoconus or were keratoconus suspects; were one-eyed patients; had undergone previous ocular surgery; had a history of herpes zoster ophthalmicus or herpes simplex keratitis; had a history of steroid-responsive rise in intraocular pressure or had a preoperative intraocular pressure of more than 21 mmHg in either eye; had diabetes mellitus, auto-immune disease, severe dry eye, connective tissue disease or significant atopy; on chronic systemic corticosteroid or immunosuppressive therapy; had a cornea thickness which would have resulted in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively or had a central corneal endothelial cell count of less than 1500 cells/mm2 in either eye

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-11; Study Completion 2005-08

PRIMARY OUTCOMES:
Comparing the efficacy, predictability, stability and safety of LASIK versus PRK

SECONDARY OUTCOMES:
Comparing wavefront aberrometry of LASIK vs PRK
Comparing patient satisfaction of LASIK vs PRK
Comparing effects of LASIK vs PRK in terms of post-surgery performance in the military setting

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, FAMS, Principal Investigator — Singapore Eye Research Institute; Benjamin Seet, Principal Investigator — Singapore Armed Forces
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore